CLINICAL TRIAL: NCT00407992
Title: An Italian, Randomized, Single-centre, Open-label Study of Occipital Nerve Stimulation in the Treatment of Chronic Migraine Headache
Brief Title: An Italian Randomized Open-label Study of Occipital Nerve Stimulation in the Treatment of Chronic Migraine Headache
Acronym: Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MFGGL113006
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Headache, Migraine
Keywords: Headache; Migraine
MeSH Terms: conditions — Migraine Disorders; Headache

ARMS (2):
- Occipital nerve stimulation ON (Experimental)
  Interventions: Device: Occipital nerve stimulation ON
- Occipital nerve stimulation OFF (Other)
  Interventions: Device: Occipital nerve stimulation off

INTERVENTIONS:
Device: Occipital nerve stimulation ON — Implant of an occipital nerve stimulator switched ON
  Arms: Occipital nerve stimulation ON
Device: Occipital nerve stimulation off — Implant of an occipital nerve stimulator switched OFF
  Arms: Occipital nerve stimulation OFF

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of occipital nerve stimulation treating Chronic Migraine Headache

ELIGIBILITY:
Inclusion Criteria:

* patients with migraine
* patients 18 years aged or above

Exclusion Criteria:

* patients which participated within the last 30 days or plan to participate during this study in another device or drug trial
* patients pregnant or planning on becoming pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number and the type of adverse events | Study period
Reduction of headache frequency and intensity | Study period

SECONDARY OUTCOMES:
Reduction in drug intake | Study period
Changes in QoL and interference in everyday activities | Study period

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Serra, Principal Investigator — IRCCS Sacro Cuore Don Calabria di Negrar
Locations (1):
- Ospedale Sacro Cuore - Don Calabria, Negrar, Verona, Italy

REFERENCES:
- [Result] Serra G, Marchioretto F. Occipital nerve stimulation for chronic migraine: a randomized trial. Pain Physician. 2012 May-Jun;15(3):245-53. PMID 22622909